CLINICAL TRIAL: NCT03482999
Title: Post-Market, Investigator Initiated, Retrospective, Audited Observational Case Series Assessing a Lysine-Derived Urethane Adhesive (TissuGlu® Surgical Adhesive) in Flap Surgery for Decubitus Repair
Brief Title: Case Series Assessing TissuGlu® Surgical Adhesive in Flap Surgery for Decubitus Repair
Status: Completed | Type: Observational
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-100-0025
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Decubitus Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: Standard Wound Closure with drains
- TissuGlu Surgical Adhesive: TissuGlu was used for approximation and adhesion of the flaps in conjunction with drains
  Interventions: Device: TissuGlu Surgical Adhesive

INTERVENTIONS:
Device: TissuGlu Surgical Adhesive
  Groups: TissuGlu Surgical Adhesive

SUMMARY:
To evaluate the impact of a high strength lysine-based adhesive (TissuGlu® Surgical Adhesive) on complications and revision rates in large flap surgery for decubitus repair.

DETAILED DESCRIPTION:
A total of 50 subjects undergoing flap surgery for decubitus repair at the Clinic for Plastic and Aesthetic Surgery, Hand Surgery, St. Joseph's Hospital in Hagen, Germany were included in a post-market investigator initiated, retrospective observational series study.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a procedure for decubitus repair
* be 22 years of age or older

Exclusion Criteria:

* expected flap size less than 5 sqcm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population included patients undergoing flap surgery for decubitus repair between March 2011 and July 2015. In October 2013, the investigator converted to the use of TissuGlu® Surgical Adhesive in conjunction with surgical drains as their standard of care for flap surgery for decubitus repair. The analysis was performed retrospectively on two consecutive cohort groups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03-28 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
reduce the post-operative duration of stay | 30 days
  duration
reduce the surgical revision rate | 30 days
  rate

SECONDARY OUTCOMES:
percent of patients requiring a revision | 30 days
  percent
duration of wound drainage | 30 days
  duration